CLINICAL TRIAL: NCT06503250
Title: Effectiveness and Safety of Atezolizumab and Bevacizumab Plus Transarterial Chemoembolization as Conversion Therapy Among Patients With Initially Unresectable Hepatocellular Carcinoma in Real-World Clinical Practice in China
Brief Title: A Study of Participants With Initially Unresectable Hepatocellular Carcinoma That is Treated With Atezolizumab and Bevacizumab Plus Transarterial Chemoembolization
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML45337
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Secondary data from medical records of approx 5 sites across China will be utilized. Patient identification period is between 28 Oct 2020 to 31 Dec 2023. The index date is defined as the earlier date of initiating Atezo+Bev or TACE after the initial diagnosis of unresectable HCC. Baseline period is defined as 60 days prior to the index date. Observation period is defined as the period from the index date until death, latest visit record during retrospective observation period, diagnosis of other primary cancer (except basal cell carcinoma), or 31 March 2024, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Radiation: Transarterial Chemoembolization

INTERVENTIONS:
Drug: Atezolizumab — Observational Study
  Other Names: Tecentriq
Drug: Bevacizumab — Observational Study
  Other Names: Avastin
Radiation: Transarterial Chemoembolization — Observational Study
  Other Names: TACE

SUMMARY:
This is a multicenter, retrospective, observational cohort study to describe the effectiveness and safety of Atezo+Bev plus Transarterial Chemoembolization (TACE) among adult patients with unresectable hepatocellular carcinoma (HCC) in real-world clinical practice in China. Eligible patients diagnosed with unresectable HCC initiating the Atezo+Bev and TACE between 28 October 2020 and 31 December 2023 will be included in this study.

ELIGIBILITY:
Inclusion criteria:

1. Initiating both Atezo+Bev and TACE between 28 October 2020 and 31 December 2023 regardless of sequencing, number of doses/cycles, and type of TACE
2. At least one dose of Atezo+Bev and one cycle of TACE spaced no longer than 4 weeks
3. Diagnosed with HCC and considered as unresectable by any of the below criteria:

   * Predicted insufficient future liver remnant volume (FLRV) after liver resection, OR
   * Predicted unattainable safe negative tumor margin resection, i.e., R0 resection, OR
   * "Unresectable" directly documented in the medical records

Exclusion Criteria:

1. No visit record after initiating both Atezo+Bev and TACE
2. Treated with other systemic therapy or resection against HCC
3. Diagnosed with concomitant cancer except for basal cell carcinoma
4. Advanced portal vein tumor thrombosis (PVTT) as defined by: Grade Vp 4, Cheng's Classification Type III or IV, or presence of a tumor thrombus in the main trunk of the portal vein, a portal vein branch contralateral to the primarily involved lobe, or superior mesenteric vein
5. China Liver Cancer (CNLC) Stage IIIb, or history of extrahepatic metastasis
6. Terminal-stage HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of adult patients with unresectable HCC who initiated Atezo+Bev plus TACE between 28 October 2020 and 31 December 2023 from approximately 3-5 study sites in China. Sites will be selected based on geographic representativeness, experience in clinical studies and HCC disease management.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Median Time to Real-World Progression-Free Survival (rwPFS) | up to approximately 12 months
  rwPFS is defined as time from the index date to the first evidence of clinician-assessed progressive disease (may include but are not limited to local tumor progression, disease recurrence, new metastasis, or clinical progression anchored by clinicians) or death from any cause.

SECONDARY OUTCOMES:
Median Time to Real-World Overall Survival (rwOS) | up to approximately 3 years
  rwOS is defined as time from the index date to death from any cause.
Median Time to Real-World Overall Response Rate (rwORR) | up to approximately 3 years
  rwORR is defined as the percentage of patients who achieved complete response (CR) or partial response (PR) after the initiation of both Atezo+Bev and TACE among patients with at least one response assessment result after the initiation of both Atezo+Bev and TACE, with reference to the assessment of tumor lesions within 60 days prior to the later initiation of Atezo+Bev or TACE.
Percentage of Participants with Serum Alpha-Fetoprotein (AFP) Reduction | up to approximately 4 years
  AFP reduction is defined as > 50% reduction in AFP level after 3 months (± 4 weeks) of the later initiation of Atezo+Bev or TACE.
Percentage of Participants with Prothrombin Induced by the Absence of Vitamin K or Antagonist-II (PIVKA-II) Reduction: | up to approximately 4 years
  PIVKA-II reduction is defined as > 50% reduction in PIVKA-II level after 3 months (± 4 weeks) of the later initiation of Atezo+Bev or TACE.
Percentage of Participants with Surgical Resection | up to approximately 4 years
  Conversion rate (surgical resection) is defined as the percentage of patients who underwent surgical resection of tumor among patients who completed the Atezo+Bev plus TACE treatment by the end of observation period.
Percentage of Participants with Adverse Events | up to approximately 4 years
  The adverse events of interest include liver function abnormality, renal function abnormality, hemorrhage, hypertension, hepatitis virus reactivation and immune-related adverse events.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Zhongshan Hospital Fudan University, Shanghai
  - Tianjin First Central Hospital, Tianjin
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical-trials/data-sharing/).